CLINICAL TRIAL: NCT02934542
Title: Comparison of Laparoscopic Procedures With and Without the Aid of the AutoLap System- a Robotic Camera Holder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.S.T. Medical Surgery Technology LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AL-65-006-P
Record Dates: First submitted 2016-10-05; First posted 2016-10-17 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2017-09

CONDITIONS: General Laparoscopic Surgeries
Keywords: Laparoscope holder; Colon resection; Right hemicolectomy; Left hemicolectomy; Sigmoid resection; Anti-reflux; Hiatal hernia
MeSH Terms: conditions — Hernia, Hiatal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (No Intervention): Patients in this group will undergo an elective standard laparoscopic procedure with a designated OR staff to maneuver the laparoscopic camera. The procedures will be performed according to the hospital and OR routine procedure.
- AutoLap Group (Experimental): Patients in this group will undergo a laparoscopic procedure using the AutoLap system. In this group the surgeon will use the AutoLap system to hold and control the movements of the laparoscopic camera.
  Interventions: Device: AutoLap system

INTERVENTIONS:
Device: AutoLap system
  Arms: AutoLap Group

SUMMARY:
The objective of this study is to evaluate the ability to reduce the number of OR personnel required while performing the following procedures: colon resections, cholecystectomies and anti-reflux/hiatal hernia surgery with the AutoLap system compared with the standard operation.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 18 years
2. Able to provide a written informed consent

Exclusion Criteria:

1. Pregnancy
2. Obesity (BMI >35 Kg/m2)
3. Contra-indications for performing laparoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2016-09; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Success rate in performing an operation with at least one OR person less | During surgery

SECONDARY OUTCOMES:
Duration of the operation | During surgery
Number of times the laparoscope is removed for cleaning | During surgery
Usability evaluation | Up to two days post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ivo A. M. J. Broeders, MD, Principal Investigator — Meander Medisch Centrum
Locations (1):
- Meander Medisch Centrum, Amersfoort, Netherlands

IPD SHARING:
Plan to Share IPD: No